CLINICAL TRIAL: NCT05997121
Title: Safety and Performance of the Hexanium TLIF System in the Treatment of Skeletally Mature Patients Suffering From Degenerative Disc Disease - Hexanium TLIF Study
Brief Title: Safety and Performance of the Hexanium TLIF System in the Treatment of Degenerative Disc Disease
Acronym: TLIF
Status: Recruiting | Type: Observational
Sponsor: SPINEVISION SAS (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: SV005
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Intervertebral Disc Degeneration
Keywords: Lumbar; Spine; Arthrodesis; Fusion; Stabilization; Oswestry disability index; Visual Analogue Score
MeSH Terms: conditions — Intervertebral Disc Degeneration; Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Transforaminal lumbar interbody fusion — Transforaminal Lumbar Interbody Fusion indicates a surgical approach in the lumbar spine to fuse the discal space between two vertebrae. These are joined by removing the disc and placing a cage in its place to restore the vertebral height. Screws and rods are also added to maintain the level secure while the bones fuse together.

SUMMARY:
The goal of this observational study is to confirm the safety and efficacy of the Hexanium TLIF system in the treatment of skeletally mature patients suffering from degenerative disc disease (disease that occurs when the spinal disk break down).

Part of their standard of care, participants will be questioned on their back and leg pains, their disability and if they have encountered any adverse effects since the Hexanium TLIF system implant surgery. Those data will be collected up to twenty four (24) months after the Hexanium TLIF system implant surgery.

DETAILED DESCRIPTION:
The Hexanium TLIF study is a multicentric, international, ambispective, post market clinical follow-up study. This means that either subjects already implanted with the Hexanium TLIF system (retrospective subjects) or subjects planned for treatment with the Hexanium TLIF (prospective subjects) can be enrolled in the study.

Standard of care subjects data up to twenty four (24) months post Hexanium TLIF system implant procedure will be collected; key data include back and leg Visual Analogue Score (VAS), Oswestry Disability Index (ODI) score, and adverse events.

Data will be collected at Month 2, Month 6, Month 12 and Month 24 post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient planned for Hexanium TLIF system implant or patient implant with Hexanium TLIF system (not prior to July 2021)
* Patient of 18 years old or more
* Patient has provided signed informed consent, or did not oppose to his/her data collection, per local regulation

Exclusion Criteria: contra-indication

* Infection, local to the operative site
* Signed of local inflammation
* Fever or leukocytosis
* Morbid obesity
* Pregnancy
* Paediatric cases, or patient still having general skeletal growth
* Spondylolisthesis unable to be reduced to Grade I
* Suspected or documented allergy or intolerance to metal
* Any case where the implant components selected for use would be too large or too small to achieve a successful result
* Any patient having inadequate tissue coverage over the operative site or inadequate bone stock or quality
* Any patient in which implant utilization would interfere with anatomical structures or expected physiological performance
* Prior fusion at the level to be treated
* Any case not needing a bone graft or fusion
* Any abnormality present which affects the normal process of bone remodelling including, but not limited to severe osteoporosis involving spine, bone absorption, osteopenia, primary or metastasis tumours involving the spine, active infection at the site or certain metabolic disorders affecting osteogenesis
* Any other condition which would preclude the potential benefit of spinal implant surgery, such as the presence of tumours or congenital abnormalities, fracture local to operating site, elevation of segmentation rate unexplained by other diseases, elevation of white blood count (WBC), or marked left shift in the WBC differential count
* Mental illness
* Any patient unwilling to cooperate with post-operative instructions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients eligible for treatment or already treated with the Hexanium TLIF system device will be offered to participate in the study; this applies to primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse device and/or procedure related events | Month 24
  Rate of the serious adverse events related to the study device and / or surgical implant procedure will be analyzed and compared to the state of the art.
Change of the Oswestry Disability Index (ODI) | Month 12
  ODI mean score at Month 12 will be compared to the ODI mean score at baseline.

SECONDARY OUTCOMES:
Fusion success | Month 2, month 6, month 12 and month 24
  Fusion rate will be analyzed and compared to the state of the art.
Change of the Oswestry Disability Index (ODI) | Month 2, month 6, and month 24
  Mean ODI score evolution score will be analyzed.
Change of the back and leg Visual Analogue Score (VAS) | Month 2, month 6, month 12 and month 24
  Back and leg VAS assessment will be analyzed.
Incidence of revision surgery at implant site | Month 2, month 6, month 12 and month 24
  Rate of revision surgery at implant site will be analyzed and compared to the state of the art.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Graziani, Professor, Principal Investigator — Hopital Privé Clairval
Locations (6):
- France (5):
  - Clinique du dos Terrefort, Bruges
  - Clinique Saint Charles, Lyon
  - Hopital privé Clairval, Marseille
  - CHRU Nancy, Nancy
  - Polyclinique Majorelle, Nancy
- Clinicque Générale Beaulieu, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No